CLINICAL TRIAL: NCT03071965
Title: Extension Study of NT-501 Ciliary Neurotrophic Factor (CNTF) Implant for Macular Telangiectasia (MacTel)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTMT-01/02E
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: MacTel (Macular Telangiectasia) Type 2
MeSH Terms: interventions — Ciliary Neurotrophic Factor; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants completed protocol NTMT-01. All participants received surgery to implant NT-501. All participants received ciliary neurotrophic factor (CNTF).
  Interventions: Biological: Ciliary neurotrophic factor (CNTF); Procedure: Surgery
- Cohort 2 (Experimental): Participants completed protocol NTMT-02. Participants for cohort 2 arm were either:
  * NT-501 group: included subjects who each had 1 study-eligible eye that had NT-501 implanted and a fellow eye that did not undergo any study intervention.
  * Sham group: included subjects who each had 1 study-eligible eye that underwent sham surgery and a fellow eye that did not undergo any study intervention.
  * Sham+NT-501 group: included subjects who had both eyes that were study-eligible, and had NT-501 implanted in 1 eye and underwent sham surgery in the contralateral eye.
  Interventions: Biological: Ciliary neurotrophic factor (CNTF); Procedure: Surgery

INTERVENTIONS:
Biological: Ciliary neurotrophic factor (CNTF) — The investigational product is the NT-501 encapsulated cell system, which consists of cells encapsulated within a semi-permeable polymer membrane and supportive matrices. NT-501 contains NTC-201 cells that secrete recombinant human CNTF, which were derived from genetically modified NTC-200 cells.
Procedure: Surgery — Surgery to implant device for NT-501
Procedure: Surgery — Sham surgery
  Arms: Cohort 2

SUMMARY:
This was a prospective, multicenter, single-masked, sham-controlled extension study designed to provide long-term safety and efficacy follow-up data for subjects with MacTel who had NT-501 implanted intraocularly and/or underwent sham surgery in the respective precursor study (NTMT-01 or NTMT-02).

A substudy was conducted in which subjects enrolled in study (NTMT-02), who had 1 study-eligible eye that underwent sham surgery, were offered the option to have NT-501 implanted in the same study eye. Of the 19 subjects who had 1 study-eligible eye and underwent sham surgery in the Cohort 2 precursor study (NTMT-02), 16 subjects elected to have NT-501 implanted in the same study eye during the substudy

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in the NTMT-01 or NTMT-02 protocol and received the NT-501 implant and/or underwent a Sham procedure
* Participant must be offered sufficient opportunity to review and to understand the informed consent form, agree to the form's contents, and provide written informed consent.

Exclusion Criteria:

* There are no Exclusion Criteria

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aaberg, Jr, MD, Study Chair — Neurotech Pharmaceuticals, LLC
Locations (11):
- United States (8):
  - Stein Eye Institute / David Geffen School of Medicine, Los Angeles, California
  - University of Miami-Miller School of Medicine, Bascom Palmer Eye Institute, Miami, Florida
  - Emory University School of Medicine, Dept of Ophthalmology, Emory University Eye Center, Atlanta, Georgia
  - NIH Clinical Center, Rockville, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Retina Associates of Cleveland, Inc, Cleveland, Ohio
  - University of Wisconsin-Madison, Department of Ophthalmology and Visual Sciences, Madison, Wisconsin
- Australia (3):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Lions Eye Institute, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort 1:
  Six subjects consented to the extension study, totaling six study eyes and six fellow eyes.
  Cohort 2:
  In NTMT-02, 64 subjects joined the extension study:
  NT-501 group: 15 subjects (15 study eyes, 15 fellow eyes). Sham group: 19 subjects (19 study eyes, 19 fellow eyes). Sham+NT-501 group: 30 subjects (1 implanted, 1 sham eye each). Cohort 2 included 128 eyes: 94 study eyes (45 NT-501, 49 sham) and 34 fellow eyes.
Units Other Than Participants: eyes
Groups:
- Cohort 1 - Implant Only: Participants who completed protocol NTMT-01 and had one NT-501 implant.
- Cohort 2 - Sham Only: Participants who completed protocol NTMT-02 and only had a sham surgery. Note, there is a subset of these participants who opted to receive an actual NT-501 implant during the extension study.
- Cohort 2 - NT-501 Implant: Participants who completed protocol NTMT-02 and had one NT-501 implant..
- Cohort 2 - Sham + NT-501 Implant: Participants who completed protocol NTMT-02 and had one NT-501 implant in one eye and sham surgery in the other.
Period: Overall Study
Arm/Group | Cohort 1 - Implant Only | Cohort 2 - Sham Only | Cohort 2 - NT-501 Implant | Cohort 2 - Sham + NT-501 Implant
Started | 6; 6 eyes | 19; 19 eyes | 15; 15 eyes | 30; 60 eyes
Switched to NT-501 | 0; 0 eyes | 16; 16 eyes | 0; 0 eyes | 0; 0 eyes
Retained NT-501 Throughout the Study | 6; 0 eyes | 16; 16 eyes | 14; 14 eyes | 30; 60 eyes
Completed | 6; 0 eyes | 18; 18 eyes | 13; 13 eyes | 27; 54 eyes
Not Completed | 0; 6 eyes | 1; 1 eyes | 2; 2 eyes | 3; 6 eyes
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 1
Not completed — COVID-19 | 0 | 1 | 0 | 1
Not completed — Other Health Reason | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Implant Only | Cohort 2 - Sham Only | Cohort 2 - NT-501 Implant | Cohort 2 - Sham + NT-501 Implant | Total
Number analyzed (Participants) | 6 | 19 | 15 | 30 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 16 | 10 | 16 | 48
  >=65 years | 0 | 3 | 5 | 14 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (5.12) | 59.4 (7.61) | 59.5 (10.82) | 63.6 (8.59) | 61.4 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 9 | 20 | 44
  Male | 2 | 8 | 6 | 10 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 18 | 14 | 29 | 67
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 4 | 16 | 11 | 28 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Ellipsoid Zone (Area of IS/OS Loss) - Cohort 1
Description: Change from baseline to 72, 84, 96 and 108 months post-surgery (based on participants' original implant date during precursor study) by SD-OCT for Cohort 1
Time Frame: 72, 84, 96, and 108 months (based on participants' original implant date during precursor study)
Population: All enrolled participants by eye
Measure: Mean (Standard Deviation); unit: mm2
Units Other Than Participants: eyes
Groups:
- Cohort 1 - Fellow Eye: Cohort 1 - Previous NTMT-01 participant's fellow untreated eye
- Cohort 1 - NT-501 Implant: Cohort 1 - Previous NTMT-01 participant's NT-501 implant eye
Arm/Group | Cohort 1 - Fellow Eye | Cohort 1 - NT-501 Implant
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
mm2
  Baseline | 0.697 (0.8334) | 0.629 (0.08135)
  72 Months Post-Surgery Actual: number analyzed (Participants) | 5 | 6
  72 Months Post-Surgery Actual: number analyzed (eyes) | 5 | 6
  72 Months Post-Surgery Actual | 1.37 (1.4648) | 1.137 (1.2905)
  72 Months Post-Surgery Change from Baseline: number analyzed (Participants) | 5 | 6
  72 Months Post-Surgery Change from Baseline: number analyzed (eyes) | 5 | 6
  72 Months Post-Surgery Change from Baseline | 0.620 (0.7526) | 0.508 (0.6348)
  84 Months Post-Surgery Actual: number analyzed (Participants) | 5 | 6
  84 Months Post-Surgery Actual: number analyzed (eyes) | 5 | 6
  84 Months Post-Surgery Actual | 1.241 (1.4691) | 1.132 (1.1194)
  84 Months Post-Surgery Change from Baseline: number analyzed (Participants) | 5 | 6
  84 Months Post-Surgery Change from Baseline: number analyzed (eyes) | 5 | 6
  84 Months Post-Surgery Change from Baseline | 0.705 (0.7474) | 0.503 (0.5001)
  96 Months Post-Surgery Actual | 1.338 (1.3264) | 1.169 (1.0987)
  96 Months Post-Surgery Change from Baseline | 0.642 (0.6922) | 0.540 (0.5159)
  108 Months Post-Surgery Actual: number analyzed (Participants) | 3 | 3
  108 Months Post-Surgery Actual: number analyzed (eyes) | 3 | 3
  108 Months Post-Surgery Actual | 0.394 (0.5156) | 0.301 (0.4909)
  108 Months Post-Surgery Change from Baseline: number analyzed (Participants) | 3 | 3
  108 Months Post-Surgery Change from Baseline: number analyzed (eyes) | 3 | 3
  108 Months Post-Surgery Change from Baseline | 0.165 (0.1558) | 0.277 (0.4605)

2. Primary Outcome: Ellipsoid Zone (Area of IS/OS Loss) - Cohort 2
Description: Change in EZ from baseline to 36, 48, 60 and 72 Months post-surgery (based on participants' original implant date during precursor study). Cohort 2 sham surgery arm includes 16 participants (16 eyes) that received an NT-501 following their Month 36 follow-up
Time Frame: Baseline to 36, 48, 60 and 72 Months post-surgery (based on participants' original implant date during precursor study)
Population: Intent to treat population by eye
Measure: Mean (Standard Error); unit: mm2
Units Other Than Participants: eyes
Groups:
- Cohort 2 - NT-501 Implant: Previous NTMT02 participant's NT-501 treated eye
- Cohort 2 - Sham: Previous NTMT-02 participant's sham surgery eye
Arm/Group | Cohort 2 - NT-501 Implant | Cohort 2 - Sham
Number analyzed (Participants) | 45 | 49
Number analyzed (eyes) | 45 | 49
mm2
  Baseline | 0.684 (0.0707) | 0.766 (0.0687)
  Change at 36 Months Post-Surgery: number analyzed (Participants) | 43 | 48
  Change at 36 Months Post-Surgery: number analyzed (eyes) | 43 | 48
  Change at 36 Months Post-Surgery | 0.259 (0.0609) | 0.279 (0.0585)
  Change at 48 Months Post-Surgery: number analyzed (Participants) | 43 | 47
  Change at 48 Months Post-Surgery: number analyzed (eyes) | 43 | 47
  Change at 48 Months Post-Surgery | 0.360 (0.0609) | 0.282 (0.0589)
  Change at 60 Months Post-Surgery: number analyzed (Participants) | 37 | 42
  Change at 60 Months Post-Surgery: number analyzed (eyes) | 37 | 42
  Change at 60 Months Post-Surgery | 0.450 (0.0644) | 0.105 (0.0760)
  Change at 72 Months Post-Surgery: number analyzed (Participants) | 27 | 32
  Change at 72 Months Post-Surgery: number analyzed (eyes) | 27 | 32
  Change at 72 Months Post-Surgery | 0.443 (0.0728) | 0.497 (0.0680)
Statistical Analysis 1: Comparison: Cohort 2 - NT-501 Implant vs Cohort 2 - Sham; Test type: Superiority; p = 0.5455, Mixed Models Analysis; Median Difference (Final Values) = -0.053, 95% CI 2-sided [-0.226 to 0.120], Standard Error of Mean 0.0881

3. Secondary Outcome: Change in Retinal Sensitivity (dB) From Baseline - Cohort 2 Only
Description: Baseline to 72 Months - analyses also presented for additional times: 36, 48, and 60 Months post-surgery (based on participants' original implant date during precursor study) . Cohort 2 sham surgery arm includes 16 participants (16 eyes) that received an NT-501 following their Month 36 follow-up in this study.
Time Frame: Baseline to 72 Months (based on participants' original implant date)
Population: Intent to Treat population by eye
Measure: Mean (Standard Error); unit: dB
Units Other Than Participants: eyes
Arm/Group | Cohort 2 - NT-501 Implant | Cohort 2 - Sham
Number analyzed (Participants) | 45 | 49
Number analyzed (eyes) | 45 | 49
dB
  Baseline | 25.688 (0.3377) | 25.672 (0.3317)
  Retinal Sensitivity Change at 36 Months Post-Surgery: number analyzed (Participants) | 43 | 45
  Retinal Sensitivity Change at 36 Months Post-Surgery: number analyzed (eyes) | 43 | 45
  Retinal Sensitivity Change at 36 Months Post-Surgery | -1.391 (0.3377) | -1.054 (0.3320)
  Retinal Sensitivity Change at 48 Months Post-Surgery: number analyzed (Participants) | 43 | 45
  Retinal Sensitivity Change at 48 Months Post-Surgery: number analyzed (eyes) | 43 | 45
  Retinal Sensitivity Change at 48 Months Post-Surgery | -2.312 (0.3376) | -1.965 (0.3319)
  Retinal Sensitivity Change at 60 Months Post-Surgery: number analyzed (Participants) | 37 | 44
  Retinal Sensitivity Change at 60 Months Post-Surgery: number analyzed (eyes) | 37 | 44
  Retinal Sensitivity Change at 60 Months Post-Surgery | -2.912 (0.3562) | -2.369 (0.3347)
  Retinal Sensitivity Change at 72 Months Post-Surgery: number analyzed (Participants) | 34 | 36
  Retinal Sensitivity Change at 72 Months Post-Surgery: number analyzed (eyes) | 34 | 36
  Retinal Sensitivity Change at 72 Months Post-Surgery | -3.047 (0.3674) | -2.909 (0.3595)

4. Secondary Outcome: Change in BCVA From Baseline for Cohort 1
Description: Baseline to 108 Months - analyses also presented for additional times: 84, 96 and 108 Months (based on participants' original implant date)
Time Frame: Baseline to 108 Months (based on participants' original implant date)
Population: Intent to Treat population by eye
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Cohort 1 - Fellow Eye | Cohort 1 - NT-501 Implant
Number analyzed (Participants) | 6 | 6
Number analyzed (eyes) | 6 | 6
letters
  Baseline Actual | 80.5 (7.34) | 75.0 (7.92)
  72 Months Post-Surgery Actual | 72.8 (11.91) | 71.8 (7.76)
  72 Months Post-Surgery Change from Baseline | -7.7 (7.23) | -3.2 (2.48)
  84 Months Post-Surgery Actual | 72.7 (9.37) | 72.3 (6.65)
  84 Months Post-Surgery Change from Baseline | -7.8 (4.83) | -2.7 (2.80)
  96 Months Post-Surgery Actual | 72.7 (8.82) | 72.3 (6.22)
  96 Months Post-Surgery Change from Baseline | -7.8 (3.43) | -2.7 (3.20)
  108 Months Post-Surgery Actual | 72.5 (8.31) | 68.8 (10.30)
  108 Months Post-Surgery Change from Baseline | -8.0 (3.74) | -6.2 (3.37)

5. Secondary Outcome: Change in BCVA From Baseline for Cohort 2
Description: Baseline to 72 Months - analyses also presented for additional times: 36, 48, and 60 Months (based on participants' original implant date during precursor study) . Cohort 2 sham surgery arm includes 16 participants (16 eyes) that received an NT-501 following their Month 36 follow-up
Time Frame: Baseline to 72 Months (based on participants' original implant date)
Population: Intent to Treat population by eye
Measure: Mean (Standard Error); unit: letters
Units Other Than Participants: eyes
Arm/Group | Cohort 2 - NT-501 Implant | Cohort 2 - Sham
Number analyzed (Participants) | 45 | 49
Number analyzed (eyes) | 45 | 49
letters
  Baseline | 77.2 (0.97) | 77.0 (0.93)
  Change at 36 Months Post-Surgery: number analyzed (Participants) | 44 | 49
  Change at 36 Months Post-Surgery: number analyzed (eyes) | 44 | 48
  Change at 36 Months Post-Surgery | -4.8 (0.80) | -3.2 (0.77)
  Change at 48 Months Post-Surgery: number analyzed (Participants) | 43 | 47
  Change at 48 Months Post-Surgery: number analyzed (eyes) | 43 | 47
  Change at 48 Months Post-Surgery | -5.7 (0.81) | -3.9 (0.78)
  Change at 60 Months Post-Surgery: number analyzed (Participants) | 41 | 45
  Change at 60 Months Post-Surgery: number analyzed (eyes) | 41 | 45
  Change at 60 Months Post-Surgery | -8.5 (0.82) | -3.9 (0.79)
  Change at 72 Months Post-Surgery: number analyzed (Participants) | 36 | 40
  Change at 72 Months Post-Surgery: number analyzed (eyes) | 36 | 40
  Change at 72 Months Post-Surgery | -10.1 (0.87) | -6.9 (0.83)

6. Secondary Outcome: Change in Reading Speed From Baseline - Cohort 2 Only
Description: Baseline to 72 Months - analyses also presented for additional times: 36, 48, and 60 Months (based on participants' original implant date during precursor study) . Cohort 2 sham surgery arm includes 16 participants (16 eyes) that received an NT-501 following their Month 36 follow-up. Note: there were
Time Frame: Baseline to 72 Months (based on participants' original implant date)
Population: Intent to Treat population by eye and based on participants who completed the reading speed assessment each timepoint
Measure: Mean (Standard Error); unit: words per minute
Units Other Than Participants: eyes
Arm/Group | Cohort 2 - NT-501 Implant | Cohort 2 - Sham
Number analyzed (Participants) | 44 | 47
Number analyzed (eyes) | 44 | 47
words per minute
  Baseline | 94.740 (6.4973) | 107.222 (6.2866)
  Reading Speed Change at 36 Months Post-Surgery: number analyzed (Participants) | 42 | 46
  Reading Speed Change at 36 Months Post-Surgery: number analyzed (eyes) | 42 | 46
  Reading Speed Change at 36 Months Post-Surgery | -8.838 (5.4428) | -17.798 (5.2686)
  Reading Speed Change at 48 Months Post-Surgery: number analyzed (Participants) | 39 | 45
  Reading Speed Change at 48 Months Post-Surgery: number analyzed (eyes) | 39 | 45
  Reading Speed Change at 48 Months Post-Surgery | -18.931 (5.5846) | -25.488 (5.3072)
  Reading Speed Change at 60 Months Post-Surgery: number analyzed (Participants) | 38 | 41
  Reading Speed Change at 60 Months Post-Surgery: number analyzed (eyes) | 38 | 41
  Reading Speed Change at 60 Months Post-Surgery | -28.627 (5.6369) | -18.324 (5.4825)
  Reading Speed Change at 72 Months Post-Surgery: number analyzed (Participants) | 33 | 38
  Reading Speed Change at 72 Months Post-Surgery: number analyzed (eyes) | 33 | 38
  Reading Speed Change at 72 Months Post-Surgery | -24.713 (5.9294) | -34.478 (5.6311)

ADVERSE EVENTS:
Time Frame: Any serious AE occurring after surgery through study completion, up to 108 months based on participants original implant date
Description: Safety Population, Serious non-ocular AEs and serious ocular AEs in the study eye
Arm/Group | Cohort 1 - Implant Only | Cohort 2 - Sham Only | Cohort 2 - NT-501 Implant | Cohort 2 - Sham + NT-501 Implant
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/19 | 1/15 | 1/30
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/19 | 4/15 | 7/30
Other Adverse Events (participants affected / at risk) | 6/6 | 18/19 | 14/15 | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Implant Only (N=6) | Cohort 2 - Sham Only (N=19) | Cohort 2 - NT-501 Implant (N=15) | Cohort 2 - Sham + NT-501 Implant (N=30)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device expulsion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Implant Only (N=6) | Cohort 2 - Sham Only (N=19) | Cohort 2 - NT-501 Implant (N=15) | Cohort 2 - Sham + NT-501 Implant (N=30)
Cataract (Eye disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Delayed dark adaptation (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Conjunctival cyst (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iris adhesions (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery embolism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subretinal fluid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital dermatitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oligodipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Artificial crown procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scar excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder suspension (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Computerised tomogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device expulsion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03071965/Prot_SAP_000.pdf